CLINICAL TRIAL: NCT05226481
Title: Investigating the Effect of Evidence-based Treatment for Post-traumatic Stress Disorder Among Youth
Status: Completed | Type: Observational
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Collaborators: Ministry of Health and Care Services, Norway (Unknown)
Responsible Party: Principal Investigator, Ane-Marthe Solheim Skar, Project leader, Norwegian Center for Violence and Traumatic Stress Studies
Other Study IDs: Implementation of TF-CBT
Record Dates: First submitted 2021-12-21; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Trauma; Mental Health Disorder; PTSD; Implementation
Keywords: TF-CBT; Trauma treatment; PTSD and Complex PTSD; Mental health organization
MeSH Terms: conditions — Wounds and Injuries; Mental Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TF-CBT: Trauma-focused cognitive-behavioral therapy (TF-CBT), an evidence-based method for the treatment of posttraumatic stress among youth, was provided to children and adolescents referred to CAMHS.
  Interventions: Other: Trauma-focused cognitive behavioral therapy (TF-CBT)

INTERVENTIONS:
Other: Trauma-focused cognitive behavioral therapy (TF-CBT) — Trauma-focused cognitive-behavioral therapy (TF-CBT) is an evidence-based method for the treatment of posttraumatic stress among youth.

SUMMARY:
Trauma-focused cognitive-behavioral therapy (TF-CBT) is an evidence-based practice (EBP) for the treatment of posttraumatic stress disorder (PTSD) and posttraumatic stress symptoms (PTSS) among children and adolescents. In the current study, data were collected from youth receiving TF-CBT in specialized child and adolescent mental health services (CAMHS) and their caregivers in 2018-2021.

DETAILED DESCRIPTION:
Implementation of TF-CBT is a state-wide initiative, funded by the Norwegian Ministry of Health and Care Services, and is without costs for the clinics and patients. The Norwegian Center for Violence and Traumatic Stress Studies (NKVTS) is responsible for the project. TF-CBT trainers at NKVTS train therapists at the participating CAMHS in TF-CBT. Data are collected to monitor the training and patient outcomes. Data are collected anonymously to support and ensure high-quality treatment and also provide the opportunity to investigate the effect of the implementation of TF-CBT in Norwegian CAMHS. In the period 2018-2021, additional data were collected as part of a larger study where the aim was to investigate the effect of the implementation leadership support on implementation outcomes (ClinicalTrials.gov Identifier: NCT03042832).

Data were collected through online questionnaires before, during, and after TF-CBT was provided based on usual care. Routine procedures for trauma exposure screening and related posttraumatic stress symptoms were implemented. Those who scored above a predefined clinical cut-off were enrolled into TF-CBT based on the child and her or his caregiver's consent.

The aim of the study is to investigate the patient outcomes and therapeutic processes in TF-CBT.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Norwegian CAMHS
* Screened for trauma exposure and PTSS

Exclusion Criteria:

* Below the age of 6 and above the age of 18

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Routine trauma and PTSS screening among children and adolescents (aged 6-18 years) referred to CAMHS.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
CATS-II (Child and Adolescent Trauma Screen, version II) | 2018-2021
  The child´s exposure to potential traumatizing events and posttraumatic stress disorder (PTSD) and complex PTSD (CPTSD) will be measured before, during, and after TF-CBT.

OTHER OUTCOMES:
Therapeutic Alliance for Youth and Caregivers (TASC) | 2018-2021
  Therapeutic alliance will be measured during and after TF-CBT.
Cognitions | 2018-2021
  Cognitions will be measured with the Child Post-Traumatic Cognitions Inventory (CPTCI)
Fidelity in TF-CBT | 2018-2021
  Audio recordings of therapy sessions will be scored for fidelity.
Life quality (EQ-5D-Y) | 2018-2021
  Life quality will be measured with the EQ-5D-Y (a child- and age-specific measure of the health-related quality of life (HRQoL)) before, during and after TF-CBT
Loneliness | 2018-2021
  Loneliness will be measured by items developed by the study group before, during and after TF-CBT.
The Client Satisfaction Questionnaire (CSQ) | 2018-2021
  Client satisfaction will be measured with the The Client Satisfaction Questionnaire (CSQ) after TF-CBT.
Pediatric Symptom Checklist (PSC) | 2018-2021
  Emotional and behavioral problems will be measured with the Pediatric Symptom Checklist (PSC) before, during and after TF-CBT

CONTACTS AND LOCATIONS:
Overall Officials: Ane-Marthe S Skar, PhD, Principal Investigator — Norwegian Center for Violence and Traumatic Stress Studies
Locations (1):
- Ane-Marthe Skar, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No